CLINICAL TRIAL: NCT04295460
Title: Effectiveness of a Dual Therapy (Dolutegravir + Lamivudine) on Reduction of the Viral Reservoir, Immune Recovery and Immune Activation Compared With a Triple Therapy (Dolutegravir + Tenofovir Alafenamide/Emtricitabine) in Treatment-naïve HIV-Infected Patients
Brief Title: Triple vs. Double Therapy in naïves HIV-Infected Patients
Acronym: TRIDUNA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Luis F. Lopez-Cortes, Principal Investigator, Hospitales Universitarios Virgen del Rocío
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIS-TAR-01-2019
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual Therapy (Experimental): Dolutegravir plus lamivudine
  Interventions: Drug: Randomize
- Triple Therapy (Active Comparator): Dolutegravir plus TAF/FTC
  Interventions: Drug: Randomize

INTERVENTIONS:
Drug: Randomize — Randomize to naive-treatment HIV-infected patients to receive dual o triple therapy as initial antiretroviral treatment
  Other Names: Triple therapy

SUMMARY:
The objective of this study is to clarify whether if starting antiretroviral treatment based on dual therapy (DTG + 3TC) could provide less control of residual HIV replication and, therefore, a detriment on immune activation and inflammation compared to starting with triple therapy, and could worsen the patients' long-term prognosis. For this purpose, the investigator has designed a randomized clinical trial where will assess the immunological recovery (CD4+/CD8+), immune activation, proliferation, senescence and apoptosis in T lymphocytes CD4+ and CD8+ cells by flow cytometry, the immune activation of monocytes/ macrophages and plasma concentrations of various inflammatory mediators by ELISAS, and the thymic function, the cellular reservoir of HIV and the degree of HIV DNA transcription by digital dropped PCR.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve HIV-1-infected patients ≥ 18 years of age.
* Plasma HIV-1 RNA >5000 and <500.000 copies/ml.
* T lymphocyte CD4+ count in peripheral blood >200/μl.
* Patients of childbearing age should consent to use a highly effective contraceptive method from 15 days before the time of inclusion of the study until 30 days after the end of it. It is considered a highly effective method:

  * Complete abstinence from penile-vaginal intercourse from 2 weeks prior to administration of Investigational Product, throughout the study, and for at least 2 weeks after discontinuation of all study medications;
  * Any intrauterine device with published data showing that the expected failure rate is <1% per year (not all intrauterine devices meet this criterion)
  * Male partner sterilization confirmed prior to the female subject's entry into the study, and this male is the sole partner for that subject.
  * Approved hormonal contraception.
  * Any other method with published data showing that the expected failure rate is <1% per year.
* Signed written informed consent prior to inclusion.

Exclusion Criteria:

* Acute HIV infection
* T lymphocyte CD4+ count in peripheral blood ≤ 200/µl
* Active opportunistic infection.
* Pregnancy at inclusion or during the follow-up
* Active hepatitis C and/or B virus co-infection.
* ALT ≥ 5 times the ULN, or ALT ≥ 3xULN and bilirubin ≥ 1.5xULN (with >35% direct bilirubin).
* Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (apart from hyperbilirubinemia or jaundice due to Gilbert's syndrome or asymptomatic gallstones).
* Subjects with severe hepatic impairment (Class C) as determined by Child-Pugh classification.
* Current or past disease that requires the use subsidiary of treatment with corticosteroids, immunomodulatory agents, interferon or chemotherapeutic agents.
* Any laboratory abnormality grade 3 or 4 according to the U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS (Annex 3)
* Concomitant use of drugs with potential major interactions with the prescribed drugs according to the respective full prescribing information.
* Estimated creatinine clearance <50ml/min.
* History or presence of allergy to the study drugs or their components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
proviral HIV-DNA | 48 and 96 weeks
  Mean changes in proviral HIV-DNA in PBMCs after 48 and 96 weeks of treatment

SECONDARY OUTCOMES:
Immune Recovery | 48 and 96 weeks
  Mean changes immune recovery assessed by CD4+/CD8+ T cell ratio.
Immune Activation | 48 and 96 weeks
  Mean changes immune activation assessed by the expression of HLA-DR and CD38 in both of CD4+ and CD8+ T cells.
Monocytes Activation | 48 and 96 weeks
  Mean changes monocytes activation (plasma sCD14 and sCD163).
Immunosenescense | 48 and 96 weeks
  Mean changes expression of markers for recent thymic emigrants (CD31), proliferation (Ki67), dysfunction (PD-1), senescence (CD57), and apoptosis (annexin A) in both CD4+ and CD8+ T cells.
Inflammation | 48 and 96 weeks
  Mean changes concentration of pro-inflammatory soluble mediator in plasma: TNF-α, IL-1β, IL-6, IP-10, IFN- γ, MIP-1α, MIP-1β, hsPCR y D-dímers.
Viral Reservoir | 48 and 96 weeks
  Mean changes viral reservoir size, evaluated by proviral HIV-DNA and HIV-RNA in peripheral blood mononuclear cells (PBMC) and CD4+ T cells isolate.

OTHER OUTCOMES:
Semen | 24 weeks
  Mean changes of HIV-RNA seminal plasma viral load
GALT | 48 weeks
  Mean changes of viral reservoir assessed as proviral HIV-DNA and HIV-RNA in GALT

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen del Rocio, Seville, Spain

REFERENCES:
- [Derived] Saborido-Alconchel A, Serna-Gallego A, Lopez-Cortes LE, Trujillo-Rodriguez M, Praena-Fernandez JM, Dominguez-Macias M, Lozano C, Munoz-Muela E, Espinosa N, Roca-Oporto C, Sotomayor C, Herrero M, Gutierrez-Valencia A, Lopez-Cortes LF. Decay kinetics of HIV-1-RNA in seminal plasma with dolutegravir/lamivudine versus dolutegravir plus emtricitabine/tenofovir alafenamide in treatment-naive people living with HIV. J Antimicrob Chemother. 2023 Sep 5;78(9):2354-2360. doi: 10.1093/jac/dkad245. PMID 37545387